CLINICAL TRIAL: NCT05697081
Title: Oral Manifestations of COVID-19 Correlated to Medical History. A Survey on Infected Medical Doctors.
Brief Title: Oral Symptoms of COVID-19 Among Infected Medical Doctors
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Eman Magdy Ahmed, Dr., Beni-Suef University
Other Study IDs: FDBSUREC/10092020/ME
Record Dates: First submitted 2023-01-20; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: COVID-19 Respiratory Infection
Keywords: COVID-19; Dysgeusia; Xerostomia
MeSH Terms: conditions — COVID-19; Dysgeusia; Xerostomia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Medical doctors infected with COVID-19 — web-based survey

SUMMARY:
Oral symptoms of corona virus disease have been reported by many studies. The lack of direct contact between the dentist and the patient during the active disease presented an obstacle to build a strong body of evidence.

the aim of the study is to report the oral symptoms of COVID-19 and correlate the occurrence of these symptoms with various disease-related factors.

DETAILED DESCRIPTION:
This is a cross-sectional web-based survey targeted Medical doctors infected with COVID-19. The survey questioned the diagnosis of the disease, the severity of the disease, the general symptoms, the oral symptoms along with drug and medical history.

The survey comprised a total of 3 main sections. The first section included demographic data and diagnostic method for COVID-19 infection. The second section included question about duration of the disease, the general manifestations of the disease, the previous medical history. History of smoking, severity of COVID-19 infection and history of hospitalization. Drug history and treatments for COVID-19. Presence of blood discrepancies during COVID-19 infection. The third section targeted detailed oral manifestations of the disease and questions about the oral hygiene and presence of previous oral lesions.

The questions about oral manifestations were designed based on a systematic search through the current literature, dated between 2019 and January 2021.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 infection
* Medical doctors

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: any medical doctors infected with COVID-19
Sampling Method: Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-29 (Actual)

PRIMARY OUTCOMES:
Occurrence of oral symptoms | 14 days of infection

CONTACTS AND LOCATIONS:
Overall Officials: Eman Magdy, Principal Investigator — Lecturer
Locations (1):
- Banī Suwayf University, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Survey